CLINICAL TRIAL: NCT02084238
Title: Safety and Efficiency Study of Low-dose IL-2 Treatment in Systemic Lupus Erythematosus
Brief Title: Low-dose IL-2( Interleukin-2) Treatment in SLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-03
Record Dates: First submitted 2014-03-08; First posted 2014-03-11 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE, IL-2
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interleukin-2 (Experimental): Interleukin-2 to treat activated SLE.
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — Patients receive low dose recombinant human Interleukin-2（HrIL-2） (1 million units every other day subcutaneously (HrIL-2 1X 106, ip, Qod) for a period of 14 days. After a 14-day rest, another cycle started) for 3-6 courses according to the situation of the disease.
  Other Names: Recombinant Human Interleukin-2,125Ala, SL Pharm

SUMMARY:
This clinical study will test the efficacy and safety of low dose IL-2 treatment in Systemic lupus erythematosus.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune syndrome affecting various organs. While available therapies, such as corticosteroids and immunosuppressive agents have improved the outcome of patients, there remains a significant unmet need for safe and more effective treatments. Dysfunction of regulatory T (Treg) cells has been detected in diverse autoimmune diseases, which can be promoted by interleukin-2 (IL-2). We hypothesized that low-dose IL-2 could be a novel therapy in active SLE patients.

This is a single center, uncontrolled, open-label study to assess the efficacy/safety of low dose IL-2 plus standard therapy in active SLE.

Methods: Each SLE patients (n=40) with Scores>=8 on the Safety of Estrogens in Lupus Erythematosus National Assessment (AELENA) version of the SLE Disease Activity Index (SLEDAI) that was refractory or relaps to glucocorticoid therapy received low-dose IL-2 (1 million units every other day subcutaneously (HrIL-2 1X 106, ip, Qod) for a period of 14 days. After a 14-day rest, another cycle started) for 3-6 cycles according to the situation of the disease. The end points were safety and clinical and immunologic response.

Expected Results: This trail will define low-dose IL-2 plus standard therapy is efficacy and safety with active lupus patients, which could be relevant to the amelioration the abnormity of T help cells in SLE patients.

ELIGIBILITY:
Inclusion Criteria:

* Meet the American College of Rheumatology criteria for the diagnosis of SLE.
* Under standard treatment (≥ 2 months) at the time of inclusion
* Background treatment failed to control flares or to permit prednisone tapering
* With at least one of the following manifestations: thrombocytopenia, disease-associated rash, mouth ulcer, non-infectious type of fever, active vasculitis, renal disorder(proteinuria>0.5g/day), neuropsychiatric SLE.
* Positive for at least one of the following laboratory tests: ANA>1:160, anti-dsDNA, immunoglobulin>20g/L, decreased C3 or C4, leukopenia<3×10^9/L, thrombocytopenia<100×10^9/L;
* SLE disease activity index(SLEDAI) ≥ 8.
* Negative HIV test.
* Negative for hepatitis B and C virus.
* Written informed consent form.

Exclusion Criteria:

* Sever chronic liver, kidney, lung or heart dysfunction; (heart failure (≥ grade III NYHA), hepatic insufficiency (transaminases> 3N) )
* Serious infection such as bacteremia, sepsis;
* Cancer or history of cancer cured for less than five years (except in situ carcinoma of the cervix or Basocellular carcinoma);
* High-dose steroid pulse therapy (>1.5mg/kg) or IV bolus of corticosteroids in the last 2 months.
* History of administration of rituximab or other biologics;
* Purified protein derivative (tuberculin) >10mm
* Mental disorder or any other chronic illness or drug-abuse that could interfere with the ability to comply with the protocol or to give information;
* Inability to comply with IL-2 treatment regimen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, MD and PhD, Principal Investigator — Peking University Institute of Rheumatology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liang K, He J, Wei Y, Zeng Q, Gong D, Qin J, Ding H, Chen Z, Zhou P, Niu P, Chen Q, Ding C, Lu L, Chen XX, Li Z, Shen N, Yu D, Deng J. Sustained low-dose interleukin-2 therapy alleviates pathogenic humoral immunity via elevating the Tfr/Tfh ratio in lupus. Clin Transl Immunology. 2021 Jun 1;10(6):e1293. doi: 10.1002/cti2.1293. eCollection 2021. PMID 34094549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2013 and May 2014,38 patients completed three cycles of recombinant human IL-2 (rhIL-2) in Dept. of Rheumatology and Immunology, Peking University People's Hospital. Patients were permitted changes in background therapy according to the treating physician's advice.
Pre-assignment Details: All the patients showed poor efficacy at least 4 weeks of stable routine treatment at the time of enrollment. Two of the enrolled patients withdrew from the study at week 8: one changed to the belimumab treatment by personal preference; the other elected changed to the cyclophosphamide treatment to reduce the frequency of hospital visits.
Groups:
- Interleukin-2: Interleukin-2 to treat activated SLE.
  Interleukin-2: Patients receive low dose recombinant human Interleukin-2（HrIL-2） (1 million units every other day subcutaneously (HrIL-2 1X 106, ip, Qod) for a period of 14 days. After a 14-day break, another cycle started) for 3-6 courses according to the situation of the disease.
Period: Overall Study
Arm/Group | Interleukin-2
Started | 40
Completed | 38
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Interleukin-2
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 31 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants] — Forty patients with active SLE were recruited; 38 patients completed three cycles of recombinant human IL-2 (rhIL-2). Two of the enrolled patients withdrew from the study at week 8: one changed to the belimumab treatment by personal preference; the other elected changed to the cyclophosphamide treatment to reduce the frequency of hospital visits.
  Participants
    Female | 36
    Male | 2
Region of Enrollment [Number; unit: partiipants] — Study location is in the Dept. of Rheumatology and Immunology, Peking University People's Hospital.
  partiipants
    China | 38
SELENA-SLEDAI score [Median (Standard Deviation); unit: score] — All patients were SLE with moderate-to-severe disease activity (Safety of Estrogens in Lupus Erythematosus National Assessment version of the Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) > 8.The total score ranges from 0 to 105 points.The higher the points values represent the worse/serious of the disease. Generally, (SELENA-SLEDAI) > 8 means the disease is moderate-to-severe active.
  score | 11.35 (3.71)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were SLE Responders (SRI)
Description: SRI response was defined as (1) a ≥ 4-point reduction in SELENA-SLEDAI score, (2) no new BILAG A score or ≤ 1 new BILAG B score, and (3) no deterioration from baseline in the physician's global assessment by ≥ 0.3 points.
Time Frame: week 2，week 4，week 6，week 8，week 10
Measure: Number; unit: participants
Groups:
- SRI Results: All 38 patients who completed therapy will be calculated the response rate at each visit time point(week 2,4,6,8,10).
Arm/Group | SRI Results
Number analyzed (Participants) | 38
participants
  Week 2 | 12
  Week4 | 27
  Week 6 | 33
  week 8 | 34
  week 10 | 34

2. Secondary Outcome: Immunological Responses
Description: Analysis regulatory CD4+ T (Treg) cells , interleukin 17 (IL-17)-producing helper T (Th17) cells and follicular helper T (Tfh) cells before and during IL-2 treatment. P values below 0.05 are considered statistically significant in this study.
Time Frame: week 0 and week 10
Population: regulatory CD4+ T (Treg) cells , interleukin 17 (IL-17)-producing helper T (Th17) cells and follicular helper T (Tfh) cells
Measure: Median (Full Range); unit: Percentage of CD4+ T cells
Groups:
- Immunological Responses 1: Treg in total CD4+T cells in 23 patients with SLE
- Immunological Responses 2: Tfh cells in CD4+ T cells in 23 patients with SLE
- Immunological Responses 3: Th17 in CD4+T cells in 23 patients with SLE
Arm/Group | Immunological Responses 1 | Immunological Responses 2 | Immunological Responses 3
Number analyzed (Participants) | 23 | 23 | 23
Percentage of CD4+ T cells
  Week 0 | 10.6 [3.54 to 17.6] | 3.93 [1.27 to 15.14] | 4.09 [1.69 to 11.18]
  Week 10 | 17.5 [4.76 to 28.2] | 2.1 [0.69 to 7.55] | 2.63 [1.24 to 7.06]
Statistical Analysis 1: Comparison: Immunological Responses 1 vs Immunological Responses 2 vs Immunological Responses 3; Comparing the data between baseline and week 10; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: The Immunologic Impact of Low Dose IL-2 Treatment in SLE Patients
Description: Laboratory measures were detected, including, C3, C4 and anti-dsDNA titres.
Time Frame: week 0 and week 10
Measure: Median (Full Range); unit: g/L
Groups:
- Laboratory Variables 1: Serum complement 3 in SLE patients
- Laboratory Variables 2: Serum complement 4 in SLE patients
- Laboratory Variables 3: Serum anti-dsDNA antibodies in patients with SLE
Arm/Group | Laboratory Variables 1 | Laboratory Variables 2 | Laboratory Variables 3
Number analyzed (Participants) | 38 | 38 | 38
g/L
  Week 0 | 0.42 [0.118 to 1.46] | 0.075 [0.017 to 0.54] | 417.9 [10 to 3987.5]
  Week 10 | 0.75 [0.45 to 1.23] | 0.157 [0.11 to 0.37] | 105.1 [17.14 to 2467.7]

4. Secondary Outcome: SELENA SLEDAI Score
Description: Assessment version of the SLE Disease Activity Index (SELENA-SLEDAI) change. The higher the score represent the worse of the disease. The total score ranges from 0 to 105 points, score> 8 means the disease is moderate-to-severe active".
Time Frame: week 0, week 10
Measure: Median (Standard Deviation); unit: score
Groups:
- SLEDAI Score: SLEDAI score at week 0 and week 10.
Arm/Group | SLEDAI Score
Number analyzed (Participants) | 38
score
  Week 0 | 11.35 (3.71)
  Week 10 | 3.775 (2.27)

5. Secondary Outcome: Number of Relapses
Description: Relapses mean that if the patient's SELENA SLEDAI Score is lower than 4 during the treatment, while the SELENA SLEDAI Score increase after stopping using the study drugs in 3 months.
Time Frame: 24 weeks
Reporting Status: Not Posted, anticipated posting 2020-04

6. Secondary Outcome: Safety Assessment
Description: Adverse events includes injection site reactions, influenza-like symptoms, infection, fever, tumor, cardiovascular event，drug-induced liver and kidney damage.
Time Frame: up to Day 180
Reporting Status: Not Posted, anticipated posting 2020-04

ADVERSE EVENTS:
Time Frame: 3 months
Description: No serious adverse events occurred.
Groups:
- IL-2 Therapy in SLE: All enrolled patients completed three cycles of recombinant human IL-2 (rhIL-2). In each cycle, 1 million IU rhIL-2 was administered subcutaneously every other day for 2 weeks, followed by a 2-week break.
Arm/Group | IL-2 Therapy in SLE
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 5/38
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IL-2 Therapy in SLE (N=38)
Injection-site reaction (Skin and subcutaneous tissue disorders) | 5 (5)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes